CLINICAL TRIAL: NCT03214731
Title: A Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Artesunate Plus Standard of Care in Active Lupus Nephritis: Pilot Study
Brief Title: Efficacy and Safety of Artesunate Plus Standard of Care in Active Lupus Nephritis
Acronym: AURORA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: The First People's Hospital of Yunnan (Other); The First Affiliated Hospital of Nanchang University (Other); General Hospital of Ningxia Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Shenzhen Second People's Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor of Medicine Director, Institute of Nephrology The First Affiliated Hospital Sun Yat-Sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AURORA
Record Dates: First submitted 2017-07-08; First posted 2017-07-12 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Lupus Nephritis
Keywords: artesunate
MeSH Terms: conditions — Lupus Nephritis | interventions — Artesunate; Reproductive Techniques, Assisted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose Art (Experimental): 25mg bid Artesunate and standard of care was given to patients
  Interventions: Drug: Artesunate
- high dose Art (Experimental): 50mg bid Artesunate and standard of care was given to patients
  Interventions: Drug: Artesunate
- placebo (Placebo Comparator): Placebo and standard of care was given to patients
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Artesunate — Artesunate was produced by pharmaceutical factory for research specifically
  Other Names: Art
  Arms: high dose Art; low dose Art
Other: placebo — placebo was produced by pharmaceutical factory for research specifically
  Arms: placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study. Study subjects are class III, IV, V, III+V, IV+V lupus nephritis patients, according to ISN/RPS 2003 classification of LN, with active lesion needing corticosteroid in combination with immunosuppressant therapy.

Subjects who meet the eligibility criteria during screening will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio: 25mg bid artesunate, 50mg bid artesunate or placebo plus standard of care (prednisone plus mycophenolate mofetil ［MMF］) for 6 month.

DETAILED DESCRIPTION:
Lupus nephritis (LN) can be observed in up to 70% of SLE patients and is often associated with a poor long-term prognosis. Artesunate, one analogues of antimalarial agent artemisinin, have immunomodulatory properties that might be useful for treating autoimmune diseases including SLE. it is still lack of solid evidence from RCT to evaluate efficacy and safety of artesunate plus standard of care in active LN. Regarding no data could be referred to decide the sample size and optimal dosage, we designed this pilot study. The result and experience of pilot study will answer these questions, and guarantee the multicenter RCT to be conducted successfully.

This is a multi-center, randomized, double-blind, placebo-controlled study. Study subjects are class III, IV, V, III+V, IV+V lupus nephritis patients, according to ISN/RPS 2003 classification of LN, with active lesion needing corticosteroid in combination with immunosuppressant therapy.

Subjects who meet the eligibility criteria during screening will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio: 25mg bid artesunate, 50mg bid artesunate or placebo plus standard of care (prednisone plus mycophenolate mofetil ［MMF］) for 6 month.

All the subjects were asked to visit the hospital for weekly follow-up for four weeks, then monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* 1, Subjects of either sex, 14-65 years of age, 2, Diagnosis of SLE according to the ACR criteria (1997), 3, Renal biopsy within 6 months prior to randomization with a histological diagnosis (ISN/RPS 2003 classification of LN) class III, IV, V, III+V and IV+V [excluding Class III(C), IV-S(C), and IV-G(C)], 4, Class IV or IV+V LN: proteinuria ≥1g/24hr (or Urinary protein: creatinine ratio≥ 1.0) or Scr>1.3mg/dl, with active urinary sediment [> 5 RBCs/hpf or> 5 WBCs/hpf (or within the reference range of the laboratory) in absence of menses and genitourinary tract infection, or presence of cellular casts (RBC or WBC casts)], 5, Class III, III+V or V LN: proteinuria ≥2g/24hr (or Urinary protein: creatinine ratio ≥ 2.0) or Scr>1.3mg/dl, 6, Provision of written informed consent by subject or guardian.

Exclusion Criteria:

1. eGFR<30ml/min/1.73m2,
2. Subjects who have previously failed both MMF (or other forms of mycophenolate) induction therapies,
3. Subjects who received an induction therapy with CTX or MMF within 3 months prior to the planned initiation of the current induction for the study,
4. Have severe active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident [CVA], cerebritis, or CNS vasculitis) requiring therapeutic intervention within 60 days of baseline (Day 0),
5. Have acute or chronic infection requiring management based on the investigator's opinion,
6. Pregnant, nursing or under unreliable contraceptive method,
7. Subjects who have been on continuous dialysis starting >2 weeks before randomization into the induction phase and/or continuous dialysis with an anticipated duration >8 weeks,
8. Have a history of kidney transplant or a plan of kidney transplant,
9. Known hypersensitivity or contraindication to any drug products or any component of these drug products they plan to receive (e.g. Artesunate, CTX, MMF, AZA, corticosteroids),
10. Have severe acute or chronic diseases (e.g. cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological or infectious diseases) which, in the opinion of the principal investigator, could confound the results of the study or put the subject at under risk,
11. Have a history of malignant neoplasm within the last 5 years, except for adequately treated carcinoma in situ of the uterine cervix,
12. Recruited by other trial and/or use study agent within 4 weeks.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Remission | 6 month
  1. Complete remission: Proteinuria < 0.3g/ 24hr, no active urinary sediment, normal albumin, stable Scr (within 15% fluctuation).
  2. Partial remission: Proteinuria between 0.3 and 2.9g /24hr and a decrease in value of at least 50% of base value, albumin≥30g/L, stable Scr (within 15% fluctuation).

CONTACTS AND LOCATIONS:
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided